CLINICAL TRIAL: NCT04920331
Title: STATUS STUDY: Pilot Open-Label Trial of Intravenous Erenumab in Patients With Status Migrainosus
Brief Title: Study of Intravenous Erenumab in Patients With Status Migrainosus
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: No Participants Enrolled
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Juliana H. VanderPluym, Principal Investigator, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 19-006424
Record Dates: First submitted 2021-06-03; First posted 2021-06-09 (Actual); Last update posted 2022-02-22 (Actual); Status verified 2022-02

CONDITIONS: Status Migrainosus
MeSH Terms: conditions — Migraine Disorders | interventions — erenumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Erenumab (Experimental): Subjects with episodes of status migrainosus will receive a single dose of IV erenumab
  Interventions: Biological: Erenumab

INTERVENTIONS:
Biological: Erenumab — 140mg single intravenous administration (60 minutes)

SUMMARY:
The investigators will evaluate the efficacy for use of intravenous erenumab 140mg for treatment of status migrainosus in an open-label, pilot study.

DETAILED DESCRIPTION:
This will be a single-center, open-label, pilot study. The investigators will enroll 15 subjects. Subjects will be recruited from the outpatient Mayo Headache Clinic. The Headache Clinic employs 5 headache specialists and 1 fellow which is sufficient staffing to support this study and recruitment of patients with status migrainosus.

Subject participation would be for a total of 28 days. Subjects will be screened at outpatient clinic visit appointments or when they call into the clinic regarding an episode of status migrainosus and interested qualified subjects will be consented and offered participation in this trial.

Once consent has been obtained, subjects will have evaluation of vital signs, pregnancy status, complete blood count, and comprehensive metabolic panel. Abnormal metabolic profile, kidney or liver function will exclude subjects. Pregnancy will exclude subjects. Qualifying subjects will be administered a single dose of intravenous erenumab at our Infusion Center at the first available appointment within 24 hours of qualifying for participation if they continue to have moderate to severe pain and monitored on-site for a minimum of 2 hours after start of drug administration.

Subjects will fill out two headache diaries following treatment. The first diary is an hourly diary with entries once every hour for 24 hours, with time point 0 defined as time of when treatment begins. Diary entry at hour 24 coincides with the time point for post-treatment day 1. Follow-up will occur by phone at post-treatment day 1. If pain and symptoms persist, patients will be directed to contact their primary headache provider to receive further management. From this point and onwards, patients will be instructed to fill out a second diary once daily for 28 consecutive calendar days following treatment. A final visit will be conducted at the end of the study at 28 days.

ELIGIBILITY:
Inclusion Criteria:

* 18 years to 70 years.
* History of migraines (with or without aura) for ≥ 12 months and history of at least 1 episode of status migrainosus based on medical records and/or patient self-report in their lifetime.
* Currently experiencing an episode of status migrainosus (non-menstrually related) per ICHD3 criteria of ≥ 3 and < 6 days.
* Migraine frequency: ≥ 2 and < 10 migraine days per month on average across the 3 months prior to screening.
* Headache (i.e., migraine and non-migraine headache) frequency: < 15 headache days per month on average across the 3 months prior to screening.
* Agree to withhold acute treatments for 24 hours after receiving erenumab IV unless medically necessary.

Exclusion Criteria:

* Older than 50 years of age at migraine onset.
* History of cluster headache or hemiplegic migraine headache.
* Past (within 4 months) or present exposure to a CGRP monoclonal antibody or CGRP small molecule receptor antagonist for migraine treatment.
* Present exposure to lasmiditan.
* New acute treatment within 7 days.
* New preventive treatment within 4 weeks.
* > 15 days acute treatment use, opioid or barbiturate use > 4 days per month.
* Use of acute treatment within 6 hours of the infusion.
* Unable to differentiate migraine from other headaches.
* Procedures (e.g., nerve blocks) or neuromodulatory devices within 7 days.
* History of major psychiatric disorder.
* History or evidence of any unstable or clinically significant medical condition, that in the opinion of the investigator, would pose a risk to subject safety or interfere with the study evaluation, procedures, or completion.
* History of myocardial infarction, stroke, transient ischemic attack, unstable angina, coronary artery bypass surgery, or other revascularization procedures within 12 months prior to screening.
* Females who are pregnant, breastfeeding, or who are trying to become pregnant.
* Not willing to use a reliable form of contraception (for women of childbearing potential) through 16 weeks after the last dose of erenumab. Acceptable methods of birth control include not having intercourse, hormonal birth control methods, intrauterine devices, surgical contraceptive methods, or two barrier methods (each partner must use a barrier method) with spermicide. A reliable form of contraception must be started prior to or at the time of starting the run-in phase. Not being of childbearing potential is defined as any woman who:
* Is post-menopausal by history, defined as:
* At least 55 years of age with cessation of menses for 12 or more months; OR
* Younger than 55 years of age but no spontaneous menses for at least 2 years; OR
* Younger than 55 years of age and spontaneous menses within the past 1 year, but currently amenorrheic (e.g., spontaneous or secondary to hysterectomy), AND with postmenopausal gonadotropin levels (luteinizing hormone and follicle-stimulating hormone levels at least 40 IU/L) or postmenopausal estradiol level (less than 5 ng/dL) or according to the definition of "postmenopausal range" for the laboratory involved; OR
* Underwent bilateral oophorectomy; OR
* Underwent hysterectomy; OR
* Underwent bilateral salpingectomy.
* Currently receiving treatment in another drug study or an investigational device study, or less than 90 days prior to screening since ending treatment on another investigational device or drug study(-ies).
* Unable to provide informed consent.
* Unlikely to be able to complete all protocol required study visits or procedures, and/or to comply with all required study procedures.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-09-07 (Actual); Primary Completion 2022-02-04 (Actual); Study Completion 2022-02-04 (Actual)

PRIMARY OUTCOMES:
Pain relief at 2 hours | 2 hours after treatment
  Number of subjects with decreased pain from moderate or severe at baseline to mild or none at 2 hours after treatment

SECONDARY OUTCOMES:
Pain freedom at 2 hours | 2 hours after treatment
  Number of subjects who become pain free at 2 hours after treatment.
Absence of most bothersome symptom at 2 hours | 2 hours after treatment
  Number of subjects with absence of most bothersome symptom at 2 hours after treatment.
Relief of most bothersome symptom at 2 hours | 2 hours after treatment
  Number of subjects with decrease in most bothersome symptom from moderate or severe at baseline to mild or none at 2 hours after treatment.
Pain freedom at 24 hours | 24 hours after treatment
  Number of subjects who become pain free at 24 hours after treatment
Pain relief at 24 hours | 24 hours after treatment
  Number of subjects with decrease in pain from moderate or severe at baseline to mild or none at 24 hours after treatment
Sustained pain freedom at 24 hours | 24 hours after treatment
  Number of subjects who are pain free at 24 hours with no use of rescue medications or relapse within 24 hours of the initial treatment.
Sustained pain freedom at 48 hours | 48 hours after treatment
  Number of subjects who are pain free at 48 hours with no use of rescue medications or relapse within 48 hours of the initial treatment.
Sustained pain relief at 24 hours | 24 hours after treatment
  Number of subjects who have pain relief at 24 hours with no use of rescue medications or relapse within 24 hours of the initial treatment.
Sustained pain relief at 48 hours | 48 hours after treatment
  Number of subjects who have pain relief at 48 hours with no use of rescue medications or relapse within 48 hours of the initial treatment.
Change in pain intensity at 2 hours | Baseline, 2 hours
  Measured using a self-reported questionnaire to rate headache pain on a numerical rating scale from 0-10, where 0 is no pain and 10 is the worst pain imaginable.
Change in pain intensity at 24 hours | Baseline, 24 hours
  Measured using a self-reported questionnaire to rate headache pain on a numerical rating scale from 0-10, where 0 is no pain and 10 is the worst pain imaginable.

CONTACTS AND LOCATIONS:
Overall Officials: Juliana VanderPluym, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Arizona, Phoenix, Arizona, United States

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials